CLINICAL TRIAL: NCT06627842
Title: OSTEOARTICULAR SEPSIS ON EQUIPMENT in Intensive Care and Continuing Care Units in France
Brief Title: OsteoArticular Sepsis in Intensive Care unitS
Acronym: OASIS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241174
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Osteoarticular Infection; Intensive Care Patients; Prosthetic Joint Infection
Keywords: Osteoarticular sepsis; sepsis; osteoarticular prothetis; intensive care; critical care; prosthetic joint infection
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Global cohort: All patients admitted to intensive care during the study period

SUMMARY:
This is an ambispective observational study of patients admitted to intensive care with a diagnosis of joint prosthesis infection (mainly knee and hip prostheses). The main objective of the study is to describe the profile, care trajectories during the stay (before or after surgery) and prognosis of patients admitted to critical care with such an infection. We also aim to compare prognosis between different groups of patients sharing the same profile and care trajectory, and to assess independent risk factors associated with 2-year mortality among the study population. Finally, we will describe the microbiological and resistance profile of severe osteoarticular device infections requiring critical care admission in France.

This is a descriptive and analytical observational study open to all French public and private hospitals.

Patient data will be retrieved prospectively from patient source files. Only 2-year data (vital status, functional data) will be collected specifically for the study, by telephone contact with the patient or his or her support person.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old.
* Hospitalization in critical care (intensive care unit or continuing care unit) between 2018 and 2022 of at least 48 hours, with prosthetic joint infection (hip, knee or shoulder prosthesis infection) as the main or associated diagnosis.

Exclusion Criteria:

* Infection on osteosynthesis material
* Infection on spinal equipment
* Patient with several infected prostheses
* Recurrence of infection on prosthesis with the same microorganism
* Patient opposing data collection
* Patient under legal protection.
* Pregnant or breast-feeding patient.
* Patient deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical care patients (intensive care and continuing care), admitted between 2018 and 2022 with a principal or associated diagnosis of prosthetic joint infection.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The profile, trajectories of care during the stay (before or after surgery) and the prognosis of patients admitted to intensive care for joint prosthesis infection over a 2-year period after admission to intensive care. | 2 years

SECONDARY OUTCOMES:
Composite endpoint reflecting poor clinical outcome | 2 years
  * Mortality, measured in critical care, at 30 days, 1 year and 2 years
  * Therapeutic failure at 2 years, defined as mechanical or septic failure.
  * Functional failure at 2 years, defined as failure to resume walking and usual activities, to return home, or to regain autonomy.
Mortality at 2 years | 2 years
Description of pathogens found in intraoperative samples, and their resistance spectrum | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carine PARE, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Lariboisière, Paris, France, France

IPD SHARING:
Plan to Share IPD: No